CLINICAL TRIAL: NCT04090697
Title: Use of Oxandrolone to Promote Growth in Infants With Hypoplastic Left Heart Syndrome: A Phase I/II Pilot Study
Brief Title: Use of Oxandrolone to Promote Growth in Infants With HLHS
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: FDA withdrawal of Oxandrin NDA and generic ANDAs
Sponsor: Carelon Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Oxandrolone
Record Dates: First submitted 2019-04-04; First posted 2019-09-16 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2023-07

CONDITIONS: Hypoplastic Left Heart; Congenital Heart Disease
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Heart Defects, Congenital | interventions — Oxandrolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxandrolone Cohort 1 (Experimental): Participants randomized to Oxandrolone Cohort 1 will receive 0.1mg/kg of oxandrolone suspended in a multi-chain triglyceride (MCT) oil buccally twice per day.
  Interventions: Drug: Oxandrolone
- Standard of Care (No Intervention): Participants randomized to standard of care will receive the standard therapies provided at the institution at which they are being treated. Control subjects will receive standard therapy with no placebo and no oxandrolone.

INTERVENTIONS:
Drug: Oxandrolone — Oxandrolone 2.5mg tabs will be suspended in multi-chain triglyceride (MCT) oil and administered buccally.
  Other Names: Anavar; Oxandrin
  Arms: Oxandrolone Cohort 1

SUMMARY:
The primary aim of this study is to determine if clinically relevant doses of buccally administered oxandrolone are safe and tolerable in neonates with hypoplastic left heart syndrome (HLHS) or other single right ventricular anomalies who have undergone a Norwood procedure. The secondary aim is to evaluate the efficacy of buccally administered oxandrolone in improving objective indices of growth and nutrition in neonates who have undergone a Norwood procedure.

DETAILED DESCRIPTION:
The proposed investigation is a Phase I/II randomized trial of 28 days of open label oxandrolone vs. no oxandrolone treatment to assess optimal dosing, safety/tolerability, and preliminary efficacy of this therapy in post-Norwood neonates with HLHS. Control subjects will receive standard therapy with no placebo and no oxandrolone.

This trial is aimed at cumulative dose finding as well as a preliminary assessment of safety/tolerability and efficacy. The design and dosing are based upon preliminary phase I data obtained as part of an ongoing protocol under IND #107706. This trial will initially include two arms (control and 0.1 mg/kg oxandrolone BID). This initial oxandrolone dose was chosen based on the preliminary data collected in the background studies conducted for this trial. There were no adverse safety outcomes in the small cohort of subjects receiving 0.1 mg/kg of oxandrolone BID.

In Cohort 1, subjects will be block randomized into each arm in a 1:4 (control to oxandrolone) ratio. An interim analysis of the safety data will be performed after the first 25 subjects in Cohort 1 have been randomized and have completed 28 days of oxandrolone therapy or observation (control group). If there are no significant differences in the primary safely/tolerability outcome and safety reviews are favorable for BID dosing, then Cohort 2 (25 subjects) will be randomized in a 1:4 ratio to the control and TID dosing arms. A similar interim analysis will be performed after Cohort 2 subjects have been randomized and completed 28 days of oxandrolone therapy. Enrollment will again be suspended during this second interim analysis to determine if dose escalation is warranted. Cohort 3A, utilizing 0.15 mg/kg oxandrolone TID would be possible if both Cohorts 1 (0.1 mg/kg BID) and 2 (0.1 mg/kg/dose TID) do not demonstrate any differences in the primary safety/tolerability outcome compared to controls and safety reviews are favorable (Figure 4). If the safety threshold is crossed, then a dose of 0.1 mg/kg/dose BID will be used for cohort 3B. An interim safety analysis will be performed after 25 subjects have been enrolled in this highest dosing arm. If at any point a risk-benefit balance in any cohort is found to be negative, then further enrollment will proceed at the lower dosing arm determined to be safe/tolerable based on the primary outcome and safety review with a 1:4 control:oxandrolone ratio and a total subject number of 100.

If the second interim safety analysis leads to the conclusion that the lower dose (0.1 mg/kg oxandrolone BID) appears to be safe and well tolerated, while the higher dose (0.1 mg/kg oxandrolone TID) is not, then the enrollment will proceed in the 0.1 mg/kg BID arm with a 1:4 ratio. If the lowest dose of oxandrolone (0.1 mg/kg BID) is found to be unsafe, then the trial will be stopped. The benefit of this approach lies in the ability to allocate patients to the highest safe dose arm thus enriching the relevance of safety/tolerability and efficacy information obtained. A higher-dose treatment arm will be used if the data reveal the initial treatment arm is not different from control with regards to the primary outcome. If no safety/tolerability effect is demonstrated, the trial will, by design, function as a randomized, controlled trial with dose-escalation. It is anticipated that the study will conclude with approximately 80 oxandrolone patients (in up to three dosing arms) and 20 control patients.

ELIGIBILITY:
Inclusion Criteria:

1. HLHS and other single ventricle of right ventricular morphology
2. Age and Norwood procedure ≤14 days of age
3. Informed consent from parent/guardian

Exclusion Criteria:

1. Small for gestational age (birth weight <10th percentile for gestational age)
2. Prematurity, defined as gestational age <37 weeks
3. Intrauterine growth retardation (birth weight ≤2.5 kg and gestational age ≥38 weeks)
4. Chromosomal abnormality, recognizable genetic syndrome or congenital anomalies of more than minor severity associated with growth failure
5. Moderate or greater right ventricular systolic dysfunction and/or moderate or greater tricuspid regurgitation prior to the Norwood procedure
6. Extracorporeal membrane oxygenation support (ECMO) prior to or within 24 hours of Norwood procedure
7. Pre-Norwood interventions (fetal intervention, balloon atrial septostomy for an intact or restrictive atrial septum)
8. Pre-Norwood pulmonary venous obstruction
9. Pre-Norwood procedure necrotizing enterocolitis and/or other gastrointestinal syndromes
10. Known contraindication to oxandrolone
11. Planned or current warfarin therapy at screening (warfarin effects are increased by anabolic drugs)
12. Significant hepatic dysfunction (elevation of serum transaminase levels greater than two times the upper limit of normal local laboratory standard at screening)
13. Hypercalcemia (>1.5 times upper normal range for lab)
14. Nephrotic syndrome
15. Unwillingness or inability to return to surgical center for follow-up evaluation
16. Participation in another clinical study that may impact growth

Max Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Biochemical evidence of hepatic dysfunction | From date of treatment initiation until the pre-SCPC evaluation or end of study participation, whichever comes first, up to 9 months
  Elevation of serum transaminase levels (alanine transaminase (ALT) and/or aspartate transaminase (AST)) >4 times the local laboratory upper limit of normal
Virilization | From date of treatment initiation until the completion of study drug therapy or end of study participation, whichever comes first, up to 28 days
  Standardized physical examination will be performed. Because there are no standard normal values for the various measurements included, each subject will serve as their own control
SAE probably or definitely related to oxandrolone therapy | From date of treatment initiation until the pre-SCPC evaluation or end of study participation, whichever comes first, up to 9 months
  Any SAE probably or definitely related to oxandrolone therapy in the opinion of the medical monitor

SECONDARY OUTCOMES:
Length-for-age z-score | At the time of completion of study drug therapy, up to 28 days after date of treatment initiation
  The efficacy of buccally administered oxandrolone will be evaluated by measuring length-for-age z-score at the end of study drug therapy
Weight-for-age z-score | At the time of completion of study drug therapy, up to 28 days after date of treatment initiation
  The efficacy of buccally administered oxandrolone will be evaluated by measuring weight-for-age z-score at the end of study drug therapy
Change in Weight-for-age z-score | From date of pre-Norwood procedure until completion of study drug therapy, up to 28 days
  The efficacy of buccally administered oxandrolone will be evaluated by measuring the change in weight-for-age z-score at the end of study drug therapy
Change in length-for-age z-score | From date of pre-Norwood procedure until completion of study drug therapy, up to 28 days
  The efficacy of buccally administered oxandrolone will be evaluated by measuring the change in length-for-age z-score at the end of study drug therapy
Prealbumin levels | During the duration of therapy
  Serum prealbumin levels will be measured weekly
Lean Body Mass | At the completion of study drug therapy, assessed up to 35 days after initiation of study drug therapy
  Lean body mass will be assessed using dual energy x-ray absorptiometry (DXA)
Decreased right ventricular systolic function | At the time of Norwood discharge and at the time of pre-SCPC evaluation, up to 9 months
  Evidence of ≥moderate right ventricular systolic dysfunction or tricuspid valve regurgitation based on qualitative assessment of clinical echocardiograms if performed

CONTACTS AND LOCATIONS:
Overall Officials: Phillip T Burch, MD, Principal Investigator — University of Mississippi Medical Center; Richard V Williams, MD, Principal Investigator — University of Utah
Locations (10):
- United States (9):
  - Children's Hospital of Atlanta, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Ann Arbor, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No